CLINICAL TRIAL: NCT06991088
Title: Research on the Cognition and Practices of Chinese Cardiologists Regarding Influenza Vaccination for Patients With Chronic Coronary Syndrome
Brief Title: Chinese Cardiologists' Knowledge/Practices on Flu Vaccine for Chronic Coronary Syndrome
Status: Not yet recruiting | Type: Observational
Sponsor: The Affiliated Hospital of Hangzhou Normal University (Other)
Responsible Party: Sponsor
Other Study IDs: AH-2025-001
Record Dates: First submitted 2025-05-19; First posted 2025-05-25 (Actual); Last update posted 2025-06-04 (Actual); Status verified 2025-05

CONDITIONS: Chinese Cardiologists
Keywords: Chronic Coronary Syndrome; Chinese Cardiologists; Knowledge Survey

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Chief Physician (Professor-level): Responses from chief physicians (professor-level) across various regions, age groups, hospital types, and years of practice in China were collected via questionnaire survey. The study assessed their knowledge level regarding influenza vaccine application in CCS patients, investigated their perceptions on whether vaccination benefits patients' health outcomes, evaluated current vaccination implementation practices, and determined their support for influenza immunization.
- Associate Chief Physician (Associate Professor-level): Responses from Associate Chief Physician (Associate Professor-level) across various regions, age groups, hospital types, and years of practice in China were collected via questionnaire survey. The study assessed their knowledge level regarding influenza vaccine application in CCS patients, investigated their perceptions on whether vaccination benefits patients' health outcomes, evaluated current vaccination implementation practices, and determined their support for influenza immunization.
- Attending Physician: Responses from Attending Physician across various regions, age groups, hospital types, and years of practice in China were collected via questionnaire survey. The study assessed their knowledge level regarding influenza vaccine application in CCS patients, investigated their perceptions on whether vaccination benefits patients' health outcomes, evaluated current vaccination implementation practices, and determined their support for influenza immunization.
- Resident Physician: Responses from chief Resident Physician across various regions, age groups, hospital types, and years of practice in China were collected via questionnaire survey. The study assessed their knowledge level regarding influenza vaccine application in CCS patients, investigated their perceptions on whether vaccination benefits patients' health outcomes, evaluated current vaccination implementation practices, and determined their support for influenza immunization.

SUMMARY:
This long-term single-center cross-sectional study evaluates physicians' knowledge of influenza vaccination in CCS patients through collected feedback, while identifying knowledge gaps and misconceptions regarding vaccination. By analyzing factors influencing physicians' recommendation practices, it provides evidence to guide future educational and policy interventions. Ultimately, the study aims to enhance cardiologists' vaccination awareness, thereby optimizing CCS patient management and reducing influenza-associated complications and mortality.

DETAILED DESCRIPTION:
This project conducts a comprehensive literature review to examine current research and practices regarding influenza vaccination for chronic coronary syndrome (CCS) patients among cardiologists worldwide. The review provides theoretical support for study design and helps identify potential causes of low vaccination rates among CCS patients in China.Based on research objectives, investigators developed a structured questionnaire covering four key dimensions:Basic demographic information、Knowledge assessment、Clinical practice patterns、Attitudes and recommendations.The survey targets cardiologists from major Chinese hospitals, employing random or stratified sampling to ensure representative sampling. Data collection will be conducted through online and offline questionnaire distribution.Statistical analysis will be performed using SPSS or equivalent software, including:Descriptive statistics、t-tests、Chi-square tests to examine how different background factors influence knowledge and practices.Findings will systematically summarize Chinese cardiologists' current understanding and behavioral patterns regarding influenza vaccination for CCS patients.

ELIGIBILITY:
Inclusion Criteria:

Cardiologists (licensed practitioners) with specialized knowledge of the association between influenza vaccination and cardiovascular diseases.

Exclusion Criteria:

* Physicians from non-cardiology specialties (e.g., surgery, general internal medicine [including respiratory and gastroenterology departments], emergency medicine).
* Physicians unable to complete the questionnaire survey.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Responses from cardiologists across various regions, age groups, professional titles, and experience levels in China, as collected in the survey.
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2025-06 (Estimated); Primary Completion 2026-07 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
cognitive status | baseline and 1-year later
  Based on a survey on "Cardiologists' Knowledge and Behavior Regarding Influenza Vaccination for Patients with Chronic Coronary Syndrome in China," regular follow-up will be conducted. The scale scores will be further improved in subsequent research.
practical situation | baseline and 1-year later
  Based on a survey on "Cardiologists' Knowledge and Behavior Regarding Influenza Vaccination for Patients with Chronic Coronary Syndrome in China," regular follow-up will be conducted. The scale scores will be further improved in subsequent research.
attitude | baseline and 1-year later
  Based on a survey on "Cardiologists' Knowledge and Behavior Regarding Influenza Vaccination for Patients with Chronic Coronary Syndrome in China," regular follow-up will be conducted. The scale scores will be further improved in subsequent research.

CONTACTS AND LOCATIONS:
Locations (1):
- MingWei Wang, Hanzhou, Zhejiang, China